CLINICAL TRIAL: NCT00380887
Title: An Open-Label, Single-Dose, Randomized, 4-Period, Partial Crossover Bioequivalence/Bioavailability Study Among Four New Formulations of Premarin 0.45 mg/Medroxyprogesterone Acetate (MPA) 1.5 mg Compared With a Reference Formulation of Premarin/MPA (Prempro) 0.45 mg/1.5 mg in Healthy Postmenopausal Women
Brief Title: Study Comparing Four New Formulations for Premarin in Healthy Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0713E1-133, 0713E1-135
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2006-09-27 (Estimated); Status verified 2006-09

CONDITIONS: Postmenopause
Keywords: bioavailability; bioequivalence; marketed product; Premarin; Medroxyprogesterone acetate; MPA; Postmenopausal; vasomotor symptoms
MeSH Terms: interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Drug: Premarin

SUMMARY:
The purpose of this study is to determine bioequivalence and bioavailability of four different Premarin/MPA test formulations versus the current formulation for Prempro.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy postmenopausal women aged 35 to 70 years
2. Nonsmoker or smoker of less than 10 cigarettes per day

Exclusion Criteria:

1. History or presence of clotting disorders
2. History or presence of cancer
3. Presence of HIV, hepatitis B or hepatitis C
4. History of drug or alcohol abuse

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer